CLINICAL TRIAL: NCT06338631
Title: Early Detection of Renal Abnormalities in Metabolically Healthy and Unhealthy Weight Excess"
Acronym: OB-KID
Status: Recruiting | Type: Observational
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Sponsor
Other Study IDs: 43C301
Record Dates: First submitted 2024-03-24; First posted 2024-03-29 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Obesity
Keywords: Metabolic phenotype; Renal function
MeSH Terms: conditions — Obesity | interventions — Diet

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adults with weight excess
  Interventions: Other: Diet

INTERVENTIONS:
Other: Diet — Pesonalized diet plan, devoloped according to Guidelines for dietary treatment of obesity, to be followed for a duration of 12 months

SUMMARY:
Overweight and obesity are increasingly prevalent worldwide. Weight excess increases the risk of in developing the metabolic syndrome, which is composed by a set of cardiometabolic risk factors such as abdominal adiposity, dyslipidemia, high blood pressure and elevated fasting glucose levels. Obesity and the metabolic syndrome are known to be risk factors for the development of chronic kidney disease. It is not clear however, whether they can be considered independent risk factors for impaired renal function and renal damage. Whereas obesity may represent an independent risk factor for renal damage, it is not clear yet if the contemporaneous presence of obesity and metabolic alterations is associated with an additional increase in the risk.

It may be important to understand the relationship between obesity, metabolic syndrome and renal health, as treatment strategies may be different for the two metabolic phenotypes of obesity, i.e., metabolically healthy obese (MHO) and metabolically unhealthy obese (MUO) patients.

The primary objective of this multicentre observational prospective study is to assess the relationship between metabolic phenotype and reduced renal function (glomerular filtration rate <90 ml/min/1.73m2 or microalbuminuria 30-300 mg/24h) in a population of 1000 patients with overweight or obesity.

The secondary aim is to study the association between diet quality, consumption of ultra-processed foods and indicators of reduced renal function and renal damage.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60 years
* BMI at least 25 kg/m2

Exclusion Criteria:

* Pregnancy or breastfeeding
* Diabetes mellitus
* Renal disease
* Systemic autoimmune diseases with possible renal involvement
* Agonistic physical activity
* Heart failure
* Pharmacologcal treatment with RAAS-inhibitors, sartans, thiazide diuretics, loop diuretics
* Urinary tract infection

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 1000 patients with weight excess or overweight (BMI > 25 kg/m2)
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Glomerular filtration rate | At baseline and after 12 months of dietary intervention programme
  Change in glomerular filtration after dietary intervention of 12 months
Microalbuminuria | At baseline and after 12 months of dietary intervention programme
  Change in microalbuminuria after dietary intervention of 12 months
Glycemia | At baseline and after 12 months of dietary intervention programme
  Change in glycemia after dietary intervention of 12 months
Body mass index | At baseline and after 12 months of dietary intervention programme
  Change in body mass index after dietary intervention of 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Istituto Auxologico Italiano, Città Studi ICANS, Milan
  - Programma Infradipartimentale di Dietoterapia nel Trapianto e nell' Insufficienza Renale Cronica, DAI di Medicina Interna ad Indirizzo Specialistico, del Policlinico Federico II di Napoli, Naples